CLINICAL TRIAL: NCT03330548
Title: Pilot Study on the Effects of a Plant-Strong Diet on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Collaborators: Rouxbe Online Culinary School (Unknown); Carl T. Hayden Medical Research Foundation (Unknown)
Responsible Party: Principal Investigator, Diane Parrington, Deputy Associate Chief of Staff for Research, Phoenix VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parrington1092
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Hyperlipidemias; Overweight and Obesity; Diabetes
Keywords: Plant-based diet; Hyperlipidemia; Diabetes; Overweight; Veterans
MeSH Terms: conditions — Hyperlipidemias; Overweight; Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 into Culinary Rx or TeleMOVE! prior to baseline measures. We plan to enroll a subset of the 80 participants to undergo a PET-MRI sub-study (total of 21 participants). This cohort requires participants to have a pooled cohort risk score of ≥ 7.5%, be willing and able to undergo FDG-PET-MRI. [The ACC/AHA pooled risk calculator utilizes information such as age, lipid profile, hypertension to estimate 10 year risk of ASCVD.
Who Masked: Outcomes Assessor
Masking Description: The assessor for the imaging studies will be blinded to the study arms of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TeleMOVE! (Active Comparator): Veterans randomized to the control arm will participate in TeleMOVE!, an arm of the Management of Overweight Veterans (MOVE!) program. TeleMOVE! is telehealth treatment program within the VA designed to improve the lives of Veterans by assisting with weight management and health promotion. This program includes daily interaction with in-home messaging technologies and clinician contact as needed
  Interventions: Behavioral: TeleMOVE!
- Culinary Rx (Experimental): Veterans randomized to the experimental arm will participate in Culinary Rx. Culinary Rx is an online instructional cooking and nutrition course that healthcare professionals can prescribe to patients who need to transition away from a Standard American Diet to a more health-supportive, whole foods, plant-based lifestyle. In partnership with The Plantrician Project, this course will focus on teaching the foundational cooking skills needed for long-term behavioral change, coupled with lifestyle education around nutrition and resources that will help users successfully face the many challenges inherent to dietary change.
  Interventions: Behavioral: Culinary Rx

INTERVENTIONS:
Behavioral: TeleMOVE! — Active comparator- telehealth treatment program for weight management and health promotion
  Arms: TeleMOVE!
Behavioral: Culinary Rx — Experimental Arm- An online instructional cooking and nutrition course to promote a whole-foods, plant-based lifestyle.
  Arms: Culinary Rx

SUMMARY:
The purpose of this study is to conduct a preliminary test of the effectiveness of various educational interventions to promote adoption of a whole-food, plant-strong diet and reduce specific cardiovascular risk factors in Veterans, and subsequently perform a preliminary pilot study on whether this dietary approach will change plaque inflammation and endothelial function.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a preliminary test of the effectiveness of various educational interventions to promote adoption of a whole-food, plant-strong diet and reduce specific cardiovascular risk factors in Veterans, and subsequently perform a preliminary pilot study on whether this dietary approach will change plaque inflammation and endothelial function. The specific aims are to conduct a preliminary examination of:

1. The feasibility of Veterans to adopt a whole-food, plant-strong diet within five weeks, following a plant-strong protocol, or within 90 days following a Plant Strong Diet (PSD) using Culinary Rx, or by TeleMOVE! (standard of care control). Feasibility factors will evaluate acceptability and practicality by a measure of the recruitment process, attrition rate, reasons for dropping, perceived benefit, and comparison of dietary pattern changes before and after the intervention.

   a. Acceptability of a plant-strong diet.
2. (Part 1) The effectiveness of a five-week whole-food, plant-strong diet on participants':

   1. Cardiovascular risk factors: Low-Density Lipoprotein, (LDL-C), High-Density Lipoprotein (HDL), Triglycerides (TG), Total Cholesterol (T Chol), C-Reactive Protein (CRP), basic chemistry panel, blood pressure, weight, waist circumference, and percent body fat.
   2. Dietary pattern, particularly the degree to which meat, fish, dairy, and added oils are decreased or eliminated from the dietary pattern; as well as the degree to which the consumption of fruits and vegetables (particularly whole-food) are increased from baseline intake, and the nutrient composition (percent of calories from protein, fat, carbohydrate, and amount of fiber) of the diet changes.
3. (Part 3) The effectiveness of completing Culinary Rx as compared to TeleMOVE! for 90 days on participants':

   1. Cardiovascular risk factors: Low-Density Lipoprotein, (LDL-C), High-Density Lipoprotein (HDL), Triglycerides (TG), Total Cholesterol (T Chol), HgbA1c, blood pressure, body mass index, weight, waist to hip ratio, and. medication usage (e.g., blood pressure, hypoglycemic, lipid lowering and anti-depressants).
   2. Dietary pattern, particularly the degree to which meat, fish, dairy, and added oils are decreased or eliminated from the dietary pattern; as well as the degree to which the consumption of fruits and vegetables (particularly whole-food) are increased from baseline intake, and the nutrient composition (percent of calories from protein, fat, carbohydrate, and amount of fiber) of the diet changes.
   3. Long-term lifestyle changes as measured by sustainability of dietary pattern and cardiovascular risk changes that occurred at 90 days and were still present at six months and one year, (excluding change in plaque inflammation and endothelial function).
4. Establish the ability of Positron Emission Tomography 18F-fluorodeoxyglucose radiopharmaceutical and magnetic resonance imaging (PET FDG-MRI) to assess serial change in plaque inflammation and plaque volume (Part 2) and then perform a pilot test to assess whether a 90-day PSD using Culinary Rx, or TeleMOVE! reduces plaque inflammation using FDG uptake on PET scan and structural changes on MRI (Part 3).

   1. Correlation analysis of aortic/carotid FDG uptake versus Framingham risk score from consecutive subjects who underwent PET FDG for clinical indications at Phoenix VA from January 1, 2010-May 31, 2015.
   2. Change in aortic/carotid plaque FDG uptake, plaque volume and aortic pulse wave velocity (measure of aortic/arterial stiffness) at baseline and following 90-day PSD using Culinary Rx, or TeleMOVE! (pilot prospective study).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: U.S. Veterans only

  1. Age >18 and < 90
  2. BMI >25 and < 40
  3. Subject has hypertension, diabetes, hyperlipidemia, or overweight/obesity based upon recognized body mass index (BMI) standards) and an interest and desire to make a lifestyle change.Ability to tolerate two FDG-PET-MRI scans.
  4. Active telephone contact information (either land line or cell phone)
  5. No contraindication to be on a PSD.
  6. Access to transportation and a functioning kitchen
  7. The ability to prepare meals independently.
  8. Access to a computer or tablet with internet access
  9. Digital camera or Smartphone

For the FDG-PET-MRI subset/portion of the study, there are additional inclusion criteria:

Inclusion criteria:

1. Pooled risk cohort score ≥ 7.5%.
2. No contraindication to magnetic resonance imaging (moderate or severe claustrophobia, ferromagnetic materials, inability to lie flat for 30 minutes).

Exclusion Criteria:

* 1. Significant unplanned weight loss within the last six months 2. BMI < 25 or > 40 3. Uncontrolled insulin-dependent diabetes with a current HbA1C of over 9% 4. Contraindication to undertake a PSD 5. Age <18 years old 6. Pregnancy/lactation 7. Taking prescribed weight loss medication(s) 8. Currently following a plant-strong diet, vegan, or medical weight loss program diet 9. Celiac disease diagnosed within the last six months 10. End-stage hepatic disease or renal disease requiring dialysis 11. Active cancer or receiving chemotherapy or radiation therapy 12. Active alcohol or substance abuse problems 13. History of eating disorders 14. Fasting triglyceride level above 350 mg/dL 15. Any psychological issues that prevent compliance 16. Unable to speak the English language 17. Have limited mobility 18. Homeless or in housing with limited kitchen access

For the FDG-PET-MRI subset/portion of the study, there are additional exclusion criteria:

1. Inability to tolerate PET scans.
2. Contraindication to magnetic resonance imaging (moderate or severe claustrophobia, ferromagnetic materials, inability to lie flat for 30 minutes)
3. Women of childbearing potential who do not have medical documentation of surgically induced menopause.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Low-density lipoprotein (LDL) | 90 days, 6 months and one year from baseline
  Fasting Low-density lipoprotein measured in milligrams per deciliter (mg/dl)

SECONDARY OUTCOMES:
Change in Dietary pattern | 90 days, 6 months and one year from baseline
  Degree to which meat, fish, dairy and added oils are decreased or eliminated from the dietary pattern; as well as the degree to which the consumption of fruits and vegetables (particularly whole-foods) are increased from baseline intake.
Change in carotid plaque | 90 days from baseline
  Plaque volume
Change in aortic pulse wave velocity | 90 days from baseline
  aortic pulse wave velocity
Change in Total Cholesterol | 90 days, 6 months and one year from baseline
  Fasting total cholesterol measured in milligrams per deciliter (mg/dl)
Change in Weight | 90 days, 6 months and one year from baseline
  Weight in kilograms measured with subject in light clothing without shoes
Change in Hemoglobin A1C (HgbA1c) | 90 days, 6 months and one year from baseline
  Hemoglobin A1c measured as %

CONTACTS AND LOCATIONS:
Overall Officials: Diane J Parrington, PhD, Principal Investigator — Phoenix VA Health Care System
Locations (1):
- Phoenix VA Health Care System, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
The study start date was before January 18, 2017, so no plan is in place.